CLINICAL TRIAL: NCT06444581
Title: Prevention of Emotional Problems in Spanish School Children Aged 8 to 12 Years Old: Evaluation of the Super Skills for Life Program
Brief Title: Effectiveness of the Universal Prevention Program Super Skills for Life in Schools
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Mireia Orgilés Amorós, Professor, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CIACIF/2021/269; CIACIF/2021/269 (Other Grant/Funding Number: Generalitat Valenciana (España))
Record Dates: First submitted 2024-05-22; First posted 2024-06-05 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Social Skills; Perfectionism; Self Esteem; Positive Affect; Negative Affect; Emotion Regulation; Depressive Symptoms; Anxiety Symptoms; Mood Disorders; Emotional Intelligence
Keywords: Social skills; Emotional skills; Prevention universal program; Program evaluation; Transdiagnostic protocol; Cognitive-behavioral protocol; Childhood; Children; School; Educational context; Group format
MeSH Terms: conditions — Social Skills; Emotional Regulation; Depression; Anxiety Disorders; Mood Disorders

STUDY DESIGN:
Intervention Model Description: Participants who meet the inclusion criteria and undergo the full baseline assessment will be assigned to the intervention group condition or to the wait-list control (WLC) group. Children assigned to the intervention condition will receive the twelve-week intervention. Participants in the WLC group will not receive any psychological intervention during the twelve-week program. Children and parents in all groups will complete the same set of measures at approximately the same time (pre-test and post-twelve weeks). Children in the WLC group will receive the intervention after the follow-up visit is completed.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group experimental (Experimental): Super Skills intervention group: multimedia material version
  The Super Skills program will be administered following the manual of the intervention by a trained therapist, as described in the section of intervention/ treatment and will be enriched with multimedia material that the implementer will project at various moments of the sessions.
  Super Skills Structured and manualized intervention with a manual for the therapist and a workbook for the children. The intervention will be administered by Super Skills-trained clinical psychologists. Sessions will take place once a week for twelve weeks, with each session lasting approximately fifty minutes. The program includes emotional education and social skills training. These contents are learned through playful exercises, activities, readings and role-playing. The intervention modality will be face-to-face.
  Interventions: Behavioral: Super Skills Schools
- Group without any intervention (No Intervention): Participants in the wait-list group will receive no psychological intervention during the twelve-week duration of the Super Skills program. Families will be informed that children in this group will receive the intervention once the posttest is completed.

INTERVENTIONS:
Behavioral: Super Skills Schools — Super Skills Structured and manualized intervention with a manual for the therapist and a workbook for the children. The intervention will be administered by Super Skills-trained clinical psychologists. Sessions will take place once a week for twelve weeks, with each session lasting approximately fifty minutes. The program includes emotional education and social skills training. These contents are learned through playful exercises, activities, readings and role-playing. The intervention modality will be face-to-face.
  Arms: Group experimental

SUMMARY:
This study aims to evaluate the effectiveness of a 12-session cognitive-behavioral transdiagnostic protocol for Spanish children aged 8 to 12 within an educational context, Super Skills for Life. The program, designed to enhance emotional management and social interaction skills, will be delivered in a group format and supplemented with multimedia materials. The study will compare outcomes between an intervention group and a wait-list control group.

DETAILED DESCRIPTION:
A 2 x 4 factorial design will be employed, with the intervention condition (intervention or waiting list) as the intergroup factor and the evaluation phase (pretest, posttest, 6-month follow-up, and 12-month follow-up) as the intragroup factor. Both parents and children will complete the same assessments at baseline, post-treatment, and follow-up stages. The researchers will analyze the changes in emotional and social variables from pre- to post-assessment in children who participate in the program.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8 to 12 years.
* Be Spanish-speaking.
* Accepting informed consent to participate in the study.

Exclusion Criteria:

* Intellectual disability, behavioral symptoms or autistic spectrum symptoms whose severity prevented the continuation of treatment.
* Current psychological or pharmacological treatment for anxiety and/or depression.
* Not accepting or revoking informed consent to participate in the study.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1100 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Social Skills Questionnaire (SSQ) (Pupil Version) | Baseline
  SSQ (Pupil Version) is a social skills assessment measure that focuses on a wide range of social behaviors in children aged 8-18. Scoring the Social Skills Questionnaire (Youth): Scores are rated from 0 (Not true), through 1 (Sometimes true), to 2 (Mostly true). The total score is computed by adding up the scores (0, 1, 2) for each item. Total scores range from 0 to 60. Higher scores on this scale indicate higher social skills in children.
Social Skills Questionnaire (SSQ) (Pupil Version) | Immediately after the intervention
  SSQ (Pupil Version) is a social skills assessment measure that focuses on a wide range of social behaviors in children aged 8-18. Scoring the Social Skills Questionnaire (Youth): Scores are rated from 0 (Not true), through 1 (Sometimes true), to 2 (Mostly true). The total score is computed by adding up the scores (0, 1, 2) for each item. Total scores range from 0 to 60. Higher scores on this scale indicate higher social skills in children.
Social Skills Questionnaire (SSQ) (Pupil Version) | 6 months after the intervention
  SSQ (Pupil Version) is a social skills assessment measure that focuses on a wide range of social behaviors in children aged 8-18. Scoring the Social Skills Questionnaire (Youth): Scores are rated from 0 (Not true), through 1 (Sometimes true), to 2 (Mostly true). The total score is computed by adding up the scores (0, 1, 2) for each item. Total scores range from 0 to 60. Higher scores on this scale indicate higher social skills in children.
Social Skills Questionnaire (SSQ) (Pupil Version) | 12 months after the intervention
  SSQ (Pupil Version) is a social skills assessment measure that focuses on a wide range of social behaviors in children aged 8-18. Scoring the Social Skills Questionnaire (Youth): Scores are rated from 0 (Not true), through 1 (Sometimes true), to 2 (Mostly true). The total score is computed by adding up the scores (0, 1, 2) for each item. Total scores range from 0 to 60. Higher scores on this scale indicate higher social skills in children.
The Positive and Negative Affect Schedule for Children-Short Form (PANAS-C-SF) | Baseline
  PANAS-C-SF assesses two subscales in children aged 6 to 18 years: positive affect (joyful, lively, happy, energetic, and proud) and negative affect (angry, fearful/scared, afraid, and sad). Responses are rated on a 5-point Likert scale ranging from 1 (very slightly or never) to 5 (very much).
The Positive and Negative Affect Schedule for Children-Short Form (PANAS-C-SF) | Immediately after the intervention
  PANAS-C-SF assesses two subscales in children aged 6 to 18 years: positive affect (joyful, lively, happy, energetic, and proud) and negative affect (angry, fearful/scared, afraid, and sad). Responses are rated on a 5-point Likert scale ranging from 1 (very slightly or never) to 5 (very much).
The Positive and Negative Affect Schedule for Children-Short Form (PANAS-C-SF) | 6 months after the intervention
  PANAS-C-SF assesses two subscales in children aged 6 to 18 years: positive affect (joyful, lively, happy, energetic, and proud) and negative affect (angry, fearful/scared, afraid, and sad). Responses are rated on a 5-point Likert scale ranging from 1 (very slightly or never) to 5 (very much).
The Positive and Negative Affect Schedule for Children-Short Form (PANAS-C-SF) | 12 months after the intervention
  PANAS-C-SF assesses two subscales in children aged 6 to 18 years: positive affect (joyful, lively, happy, energetic, and proud) and negative affect (angry, fearful/scared, afraid, and sad). Responses are rated on a 5-point Likert scale ranging from 1 (very slightly or never) to 5 (very much).
Measured by the Cognitive Emotion Regulation Questionnaire (CERQ-k) | Baseline
  CERQ-k consists of 36 items that measure nine cognitive coping strategies. Each subscale represents one cognitive coping strategy: Self-blame, Other blame, Acceptance, Planning, Positive refocusing, Rumination or focus on thought, Positive reappraisal, Putting into perspective, and Catastrophizing. The response format of the items is a five-point scale from (almost) never to (almost) always. Each item is rated 1 to 5 points. Minimum value 36 and maximum value 180.
Measured by the Cognitive Emotion Regulation Questionnaire (CERQ-k) | Immediately after the intervention
  CERQ-k consists of 36 items that measure nine cognitive coping strategies. Each subscale represents one cognitive coping strategy: Self-blame, Other blame, Acceptance, Planning, Positive refocusing, Rumination or focus on thought, Positive reappraisal, Putting into perspective, and Catastrophizing. The response format of the items is a five-point scale from (almost) never to (almost) always. Each item is rated 1 to 5 points. Minimum value 36 and maximum value 180.
Measured by the Cognitive Emotion Regulation Questionnaire (CERQ-k) | 6 months after the intervention
  CERQ-k consists of 36 items that measure nine cognitive coping strategies. Each subscale represents one cognitive coping strategy: Self-blame, Other blame, Acceptance, Planning, Positive refocusing, Rumination or focus on thought, Positive reappraisal, Putting into perspective, and Catastrophizing. The response format of the items is a five-point scale from (almost) never to (almost) always. Each item is rated 1 to 5 points. Minimum value 36 and maximum value 180.
Measured by the Cognitive Emotion Regulation Questionnaire (CERQ-k) | 12 months after the intervention
  CERQ-k consists of 36 items that measure nine cognitive coping strategies. Each subscale represents one cognitive coping strategy: Self-blame, Other blame, Acceptance, Planning, Positive refocusing, Rumination or focus on thought, Positive reappraisal, Putting into perspective, and Catastrophizing. The response format of the items is a five-point scale from (almost) never to (almost) always. Each item is rated 1 to 5 points. Minimum value 36 and maximum value 180.
Baseline children's reported anxiety symptoms. Measured by Spence Children's Anxiety Scale Child Report Short (SCAS-C-8) | Baseline
  SCAS-C-8 measures symptoms severity of the DSMIV anxiety disorders in children. Symptom frequency is recorded on a 3-point Likert scale from 0 (never) to 3 (always). This yields a minimum possible score of 0 and a maximum possible score of 24. Higher scores indicating greater severity of symptoms.
Baseline children's reported anxiety symptoms. Measured by Spence Children's Anxiety Scale Child Report Short (SCAS-C-8) | Immediately after the intervention
  SCAS-C-8 measures symptoms severity of the DSMIV anxiety disorders in children. Symptom frequency is recorded on a 3-point Likert scale from 0 (never) to 3 (always). This yields a minimum possible score of 0 and a maximum possible score of 24. Higher scores indicating greater severity of symptoms.
Baseline children's reported anxiety symptoms. Measured by Spence Children's Anxiety Scale Child Report Short (SCAS-C-8) | 6 months after the intervention
  SCAS-C-8 measures symptoms severity of the DSMIV anxiety disorders in children. Symptom frequency is recorded on a 3-point Likert scale from 0 (never) to 3 (always). This yields a minimum possible score of 0 and a maximum possible score of 24. Higher scores indicating greater severity of symptoms.
Baseline children's reported anxiety symptoms. Measured by Spence Children's Anxiety Scale Child Report Short (SCAS-C-8) | 12 months after the intervention
  SCAS-C-8 measures symptoms severity of the DSMIV anxiety disorders in children. Symptom frequency is recorded on a 3-point Likert scale from 0 (never) to 3 (always). This yields a minimum possible score of 0 and a maximum possible score of 24. Higher scores indicating greater severity of symptoms.
Measured by Mood and Feelings Questionnaire - Short Version (MFQS) | Baseline
  It assess depressive symptoms experienced in the past two weeks. The MFQS provides an overall score (minimum value 0, maximum value 26). Higher scores indicate more severe symptoms.
Measured by Mood and Feelings Questionnaire - Short Version (MFQS) | Immediately after the intervention
  It assess depressive symptoms experienced in the past two weeks. The MFQS provides an overall score (minimum value 0, maximum value 26). Higher scores indicate more severe symptoms.
Measured by Mood and Feelings Questionnaire - Short Version (MFQS) | 6 months after the intervention
  It assess depressive symptoms experienced in the past two weeks. The MFQS provides an overall score (minimum value 0, maximum value 26). Higher scores indicate more severe symptoms.
Measured by Mood and Feelings Questionnaire - Short Version (MFQS) | 12 months after the intervention
  It assess depressive symptoms experienced in the past two weeks. The MFQS provides an overall score (minimum value 0, maximum value 26). Higher scores indicate more severe symptoms.
Baseline level of physical and emotional well-being reported by children as measured by the KidKINDL_children questionnaire. | Baseline
  The KidKINDL_children measures assess physical and emotional well-being of children aged 7 to 13 years across six dimensions: physical well-being, psychological well-being, self-esteem, family, social relationships, and school. Children rate each item on a 5-point Likert scale: never (1), almost never (2), sometimes (3), almost always (4), and always (5). The total score is calculated by adding the scores for each dimension (range for each dimension: 4 to 20 points). Higher scores on each subscale and on the total scale indicate lower symptoms in children.
Level of physical and emotional well-being reported by children as measured by the KidKINDL_children questionnaire. | Immediately after the intervention
  The KidKINDL_children measures assess physical and emotional well-being of children aged 7 to 13 years across six dimensions: physical well-being, psychological well-being, self-esteem, family, social relationships, and school. Children rate each item on a 5-point Likert scale: never (1), almost never (2), sometimes (3), almost always (4), and always (5). The total score is calculated by adding the scores for each dimension (range for each dimension: 4 to 20 points). Higher scores on each subscale and on the total scale indicate lower symptoms in children.
Level of physical and emotional well-being reported by children as measured by the KidKINDL_children questionnaire. | 6 months after the intervention
  The KidKINDL_children measures assess physical and emotional well-being of children aged 7 to 13 years across six dimensions: physical well-being, psychological well-being, self-esteem, family, social relationships, and school. Children rate each item on a 5-point Likert scale: never (1), almost never (2), sometimes (3), almost always (4), and always (5). The total score is calculated by adding the scores for each dimension (range for each dimension: 4 to 20 points). Higher scores on each subscale and on the total scale indicate lower symptoms in children.
Level of physical and emotional well-being reported by children as measured by the KidKINDL_children questionnaire. | 12 months after the intervention
  The KidKINDL_children measures assess physical and emotional well-being of children aged 7 to 13 years across six dimensions: physical well-being, psychological well-being, self-esteem, family, social relationships, and school. Children rate each item on a 5-point Likert scale: never (1), almost never (2), sometimes (3), almost always (4), and always (5). The total score is calculated by adding the scores for each dimension (range for each dimension: 4 to 20 points). Higher scores on each subscale and on the total scale indicate lower symptoms in children.
Self-Concept Form 5 (AF-5) | Baseline
  It measures global satisfaction with self-concept (minimum value 0 and maximum value 120) and five dimensions (minimum value 0 and maximum value 24): Social (performance in social relationships); Academic/Professional (student/worker role); Emotional (perception of emotional state in general and in specific situations); Family (participation and integration into the family unit); and Physical self-concept (appearance and physical condition). Higher scores indicate greater satisfaction with self-image.
Self-Concept Form 5 (AF-5) | Immediately after the intervention
  It measures global satisfaction with self-concept (minimum value 0 and maximum value 120) and five dimensions (minimum value 0 and maximum value 24): Social (performance in social relationships); Academic/Professional (student/worker role); Emotional (perception of emotional state in general and in specific situations); Family (participation and integration into the family unit); and Physical self-concept (appearance and physical condition). Higher scores indicate greater satisfaction with self-image.
Self-Concept Form 5 (AF-5) | 6 months after the intervention
  It measures global satisfaction with self-concept (minimum value 0 and maximum value 120) and five dimensions (minimum value 0 and maximum value 24): Social (performance in social relationships); Academic/Professional (student/worker role); Emotional (perception of emotional state in general and in specific situations); Family (participation and integration into the family unit); and Physical self-concept (appearance and physical condition). Higher scores indicate greater satisfaction with self-image.
Self-Concept Form 5 (AF-5) | 12 months after the intervention
  It measures global satisfaction with self-concept (minimum value 0 and maximum value 120) and five dimensions (minimum value 0 and maximum value 24): Social (performance in social relationships); Academic/Professional (student/worker role); Emotional (perception of emotional state in general and in specific situations); Family (participation and integration into the family unit); and Physical self-concept (appearance and physical condition). Higher scores indicate greater satisfaction with self-image.

SECONDARY OUTCOMES:
The Child-Adolescent Perfectionism Scale (CAPS-S) | Baseline
  CAPS-S is an instrument designed to assess perfectionism in a Spanish child population aged between 8 and 11. It includes 13 items structured into 3 factors: Self-Oriented Perfectionism-Striving (SOP-Striving), Self-Oriented Perfectionism-Critical (SOP-Critical), and Socially Prescribed Perfectionism (SPP). Items are rated using a 5-point scale ranging from 1 (False - Not at all true of me) to 5 (Very True of me). Higher scores on this scale indicate higher levels of perfectionism in children.
The Child-Adolescent Perfectionism Scale (CAPS-S) | Immediately after the intervention
  CAPS-S is an instrument designed to assess perfectionism in a Spanish child population aged between 8 and 11. It includes 13 items structured into 3 factors: Self-Oriented Perfectionism-Striving (SOP-Striving), Self-Oriented Perfectionism-Critical (SOP-Critical), and Socially Prescribed Perfectionism (SPP). Items are rated using a 5-point scale ranging from 1 (False - Not at all true of me) to 5 (Very True of me). Higher scores on this scale indicate higher levels of perfectionism in children.
The Child-Adolescent Perfectionism Scale (CAPS-S) | 6 months after the intervention
  CAPS-S is an instrument designed to assess perfectionism in a Spanish child population aged between 8 and 11. It includes 13 items structured into 3 factors: Self-Oriented Perfectionism-Striving (SOP-Striving), Self-Oriented Perfectionism-Critical (SOP-Critical), and Socially Prescribed Perfectionism (SPP). Items are rated using a 5-point scale ranging from 1 (False - Not at all true of me) to 5 (Very True of me). Higher scores on this scale indicate higher levels of perfectionism in children.
The Child-Adolescent Perfectionism Scale (CAPS-S) | 12 months after the intervention
  CAPS-S is an instrument designed to assess perfectionism in a Spanish child population aged between 8 and 11. It includes 13 items structured into 3 factors: Self-Oriented Perfectionism-Striving (SOP-Striving), Self-Oriented Perfectionism-Critical (SOP-Critical), and Socially Prescribed Perfectionism (SPP). Items are rated using a 5-point scale ranging from 1 (False - Not at all true of me) to 5 (Very True of me). Higher scores on this scale indicate higher levels of perfectionism in children.
Baseline level of physical and emotional well-being reported by parents as measured by the Kid_KiddoKINDL-R questionnaire | Baseline
  The Kid_KiddoKINDL-R measures assess physical and emotional well-being of children aged 7 to 17 years across six dimensions: physical well-being, psychological well-being, self-esteem, family, social relationships, and school. Parents rate each item on a 5-point Likert scale: never (1), almost never (2), sometimes (3), almost always (4), and always (5). The total score is calculated by adding the scores for each dimension (range for each dimension: 4 to 20 points). Higher scores on each subscale and on the total scale indicate lower symptoms in children
Level of physical and emotional well-being reported by parents immediately after the intervention measured by the Kid_KiddoKINDL-R questionnaire | Immediately after the intervention
  The Kid_KiddoKINDL-R measures assess physical and emotional well-being of children aged 7 to 17 years across six dimensions: physical well-being, psychological well-being, self-esteem, family, social relationships, and school. Parents rate each item on a 5-point Likert scale: never (1), almost never (2), sometimes (3), almost always (4), and always (5). The total score is calculated by adding the scores for each dimension (range for each dimension: 4 to 20 points). Higher scores on each subscale and on the total scale indicate lower symptoms in children
Level of physical and emotional well-being reported by parents 6 months after the intervention measured by the Kid_KiddoKINDL-R questionnaire | 6 months after the intervention
  The Kid_KiddoKINDL-R measures assess physical and emotional well-being of children aged 7 to 17 years across six dimensions: physical well-being, psychological well-being, self-esteem, family, social relationships, and school. Parents rate each item on a 5-point Likert scale: never (1), almost never (2), sometimes (3), almost always (4), and always (5). The total score is calculated by adding the scores for each dimension (range for each dimension: 4 to 20 points). Higher scores on each subscale and on the total scale indicate lower symptoms in children
. Level of physical and emotional well-being reported by parents at 12 months measured by the Kid_KiddoKINDL-R questionnaire | 12 months after the intervention
  The Kid_KiddoKINDL-R measures assess physical and emotional well-being of children aged 7 to 17 years across six dimensions: physical well-being, psychological well-being, self-esteem, family, social relationships, and school. Parents rate each item on a 5-point Likert scale: never (1), almost never (2), sometimes (3), almost always (4), and always (5). The total score is calculated by adding the scores for each dimension (range for each dimension: 4 to 20 points). Higher scores on each subscale and on the total scale indicate lower symptoms in children

CONTACTS AND LOCATIONS:
Overall Officials: Mireia Orgilés Amorós, professor, Study Director — Miguel Hernadez University of Elche
Locations (1):
- Department of Health Psychology. Miguel Hernandez University of Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Starting after finishing all analysis and publication.
Access Criteria: Upon request and verification by the principal investigator to consult the available data. The use of the data for distribution in any format is not permitted.

REFERENCES:
- [Result] Orgiles M, Fernandez-Martinez I, Espada JP, Morales A. Spanish version of Super Skills for Life: short- and long-term impact of a transdiagnostic prevention protocol targeting childhood anxiety and depression. Anxiety Stress Coping. 2019 Nov;32(6):694-710. doi: 10.1080/10615806.2019.1645836. Epub 2019 Jul 23. PMID 31334667
- [Result] Fernandez-Martinez I, Orgiles M, Morales A, Espada JP, Essau CA. One-Year follow-up effects of a cognitive behavior therapy-based transdiagnostic program for emotional problems in young children: A school-based cluster-randomized controlled trial. J Affect Disord. 2020 Feb 1;262:258-266. doi: 10.1016/j.jad.2019.11.002. Epub 2019 Nov 4. PMID 31733917
- [Result] Melero S, Morales A, Espada JP, Mendez X, Orgiles M. Effectiveness of Group vs. Individual Therapy to Decrease Peer Problems and Increase Prosociality in Children. Int J Environ Res Public Health. 2021 Apr 9;18(8):3950. doi: 10.3390/ijerph18083950. PMID 33918640
- [Result] Essau CA, Sasagawa S, Jones G, Fernandes B, Ollendick TH. Evaluating the real-world effectiveness of a cognitive behavior therapy-based transdiagnostic program for emotional problems in children in a regular school setting. J Affect Disord. 2019 Jun 15;253:357-365. doi: 10.1016/j.jad.2019.04.036. Epub 2019 Apr 16. PMID 31078836
- [Result] Yoga Ratnam KK, Nik Farid ND, Yakub NA, Dahlui M. The Effectiveness of the Super Skills for Life (SSL) Programme in Promoting Mental Wellbeing among Institutionalised Adolescents in Malaysia: An Interventional Study. Int J Environ Res Public Health. 2022 Jul 30;19(15):9324. doi: 10.3390/ijerph19159324. PMID 35954681
- See also: The Child Research Center is the Miguel Hernández University's center dedicated to child and adolescent mental health — https://centroinvestigacioninfancia.umh.es/
- See also: Super Skills for Life program website in world — https://www.superskillsforlife.com/